CLINICAL TRIAL: NCT02890862
Title: Three-dimensional Kinematic Motion Analysis of Finger and Wrist During Daily
Brief Title: Three-dimensional Kinematic Motion Analysis of Finger and Wrist During Daily Activities
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Institute for Biomechanics, ETH Zürich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2015-0395
Record Dates: First submitted 2016-08-18; First posted 2016-09-07 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Hand Injuries
Keywords: Kinematics; Activity of Daily living; 3D motion analysis
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 20 healthy volunteers
- Dupuytren disease: 10 patients dupuytren disease
- Tendon pathology: 10 patients with tendon pathology
- wrist osteoarthritis: 10 patients with wrist osteoarthritis

SUMMARY:
Development of reliable and objective evaluation methods is required for natural upper-extremity tasks. Three-dimensional imaging measurement techniques are a powerful tool for quantitative assessment of multijoint movements.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of 20 healthy, right dominant hands
* 10 patients with tendon pathologies
* 10 patients with Dupuytren disease
* 10 patients with osteoarthritis of the wrist
* Patients older than 18 years
* Patient willing and able to give written informed consent to participate in the study

Exclusion Criteria:

* Inflammatory disease (e.g. rheumatoid arthritis)
* Pregnant women
* German language barrier to complete the questionnaires
* Any disease process that would preclude accurate evaluation (e.g. neuromuscular, psychiatric or metabolic disorder)
* Legal incompetence
* Participation in any other medical device or medicinal product study within the previous months that could influence the results of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of healty persons, patients with tendon pathologies, arthrosis and dupuytren disease. In the future the new findings should assist the decision of surgical procedures.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Joint angle of finger and wrist (Vicon) | 36 months
  Position of the Skin markers be measured with the Vicon cameras and the Joint angles will be calculated with matlab program. Maximum range of motion will be compared between first and second measurement.
Joint angle of finger and wrist (Goniometer) | 36 months
  Maximum range of motion will be compared between first and second measurement

SECONDARY OUTCOMES:
Objective functional parameters: - daily activities: open a bottle, open a glass, type 3 words, write 3 words, turn a key, pick up small object, move heavy object (1/3kg), dart-throwing motion | 36 months
  Position of the Skin markers be measured with the Vicon cameras during daily activities and the joint angles will be calculated with matlab program.
Subjective functional parameters: - Mayo Wrist Score - Krimmer Wrist Score - Short Version of the Disability of the Arm, Shoulder and Hand questionnaire (QuickDASH) | 36 months
  Mayo Wrist Score: On a scale from 0-100 points, 91-100 points is a excellent result, 81-90 a good results, 65-80 a satisfactory result and less than 65 points a poor result Krimmer Wrist Score: On a scale from 0-100 points, more than 80 is a excellent result, 65-80 a good result, 50-65 a satisfactory result and 0-50 a poor result.
  QuickDASH: At least 10 of the 11 items must be completed for a score to be calculated. The assigned values for all completed responses are simply summed and averaged, producing a score out of five. This value is then transformed to a score out of 100 by subtracting one and multiplying by 25. This transformation is done to make the score easier to compare to other measures scaled on a 0-100 scale. A higher score indicates greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Calcagni, PD Dr. med., Principal Investigator — Plastic surgery and Handsurgery USZ
Locations (1):
- University Hospital Zurich, Center for Reconstructive Surgery, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No